CLINICAL TRIAL: NCT00512356
Title: Study to Evaluate the Efficacy and Safety of Anti-Adhesion Product in the Prevention of Intraperitoneal Adhesions
Brief Title: Efficacy and Safety Study of Anti-Adhesion Product in the Prevention of Intraperitoneal Adhesions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 549902
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Intraperitoneal Adhesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Investigational product group (Experimental): Anti-Adhesion Product was applied to the rectal stump and the incision line.
  Like in the control group, surgical measures to prevent adhesions were also taken, e.g. using minimum traumatizing surgical technique, using powder-free gloves.
  Interventions: Biological: Anti-Adhesion Product
- Control group (No Intervention): Only surgical measures to prevent adhesions were taken, e.g. using minimum traumatizing surgical technique, using powder-free gloves. No specific additional treatment was applied.

INTERVENTIONS:
Biological: Anti-Adhesion Product — Anti-Adhesion Product (AAP) is a biological two-component product of human origin. The components of AAP are lyophilized Anti-Adhesion Protein Concentrate (AAPC), containing fibrinogen, lyophilized Thrombin Concentrate (TC) and the respective diluents for the reconstitution of the components.
  Arms: Investigational product group

SUMMARY:
The objective of this study was to evaluate the efficacy of the Anti-Adhesion Product (AAP) in preventing or reducing post-operative adhesion formation and re-formation in a subject population having abdominal surgery and being left with a rectal stump and a temporary stoma from a first procedure and scheduled for a laparoscopy/ laparotomy as a second procedure in the normal treatment of the subjects' disease. In both study groups, surgical measures to prevent adhesions were taken, e.g. using minimum traumatizing surgical technique, using powder-free gloves. In the investigational product group, AAP was applied to the rectal stump and the incision line while no specific additional treatment was applied in the control group. The surgeon assessed preexisting adhesions during the first surgery. Newly developed and re-formed adhesions were evaluated during the second surgery by a surgeon or assistant who did not know the result of randomization. The safety of the study drug was also monitored.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from the subject or the subject's legally authorized representative prior to study entry
* Male or female subjects > 18 years of age
* Subjects undergoing abdominal surgery with the possibility that a rectal stump would remain due to one or more of the following reasons: inflammatory bowel diseases, neoplasm, colon diverticulitis, colonic obstruction, colon polyposis, peritoneal trauma, fistula, incontinence, or other reasons
* Subjects for whom a second abdominal surgery is planned within approximately eight months of the first surgical procedure.

Exclusion Criteria:

Pre operative:

* Pregnancy and lactation period
* Subjects concurrently participating in another clinical trial with a drug or a device
* Subjects who have participated in a clinical trial with a drug or a device within 30 days prior to this study
* Subjects who have had abdominal/pelvic surgery within six months prior to this study
* Subjects who have received or will receive (approximately within the next eight months) abdominal/pelvic irradiation

Intra operative:

* Subjects with peritonitis
* Subjects with gastrointestinal metastatic cancer, or cancer growing per continuitatem into surrounding tissues
* Subjects treated with hemostatic agents (e.g. fibrin sealant, collagen, oxidized cellulose) during the first surgery
* Subjects treated with adhesion prevention agents other than the Anti-Adhesion Product (AAP) (e.g. Intergel® Adhesion Prevention Solution, Seprafilm® Membrane) during the first surgery
* Subjects with major fecal contamination needing an abdominal lavage during the first surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2000-12; Primary Completion 2003-02-25 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adhesions around the rectal stump and/or incision line

SECONDARY OUTCOMES:
Number of subjects with no adhesions
Extent and severity of adhesions around the rectal stump
Extent and severity of adhesions at the incision line
Incidence, extent and severity of adhesions at sites other than the rectal stump and incision line
Time to reach and free the rectal stump
Safety (laboratory evaluation, recording of adverse experiences)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, MD, Principal Investigator — Baxter Healthcare Corporation
Locations (7):
- Denmark (2):
  - Copenhagen University Hospital, Rigshospitalet Department of Gastroenterologic Surgery, Copenhagen
  - Odense University Hospital, Surgical Gastroenterology Department, Odense
- Poland (2):
  - Klinika Chirurgii Ogolnej Onkologicznej i Klatiki Piersiowej CSK WAM, Warsaw
  - Im. Marii Sklodowskiej-Curie, Centrum Onkologii-Instytut, Warsaw
- Sweden (3):
  - Göteborg University, Department of Surgery, Colorectal Unit, Gothenburg
  - Söder Sjukhuset, Department of Surgery, Stockholm
  - Uddevalla Sjukhus, Kirurg Kliniken, Uddevalla